CLINICAL TRIAL: NCT05734755
Title: Effects of an Individualized Dietary Behavioural Change (IDBC) Programme and Exercise Training in Combination or Separately on Managing Sarcopenic Obesity in Community-dwelling Older Adults: A Randomized Controlled Trial
Brief Title: Dietary Programme and Exercise Training in Combination or Separately on Managing Sarcopenic Obesity in Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr. Justina Liu Yat Wa, Principal Investigator, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20220722001
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Sarcopenic Obesity
Keywords: Sarcopenic Obesity; Dietary intervention; Behavioural Change; Lifestyle intervention; RCT

STUDY DESIGN:
Intervention Model Description: A four-arm RCT to evaluate the effects of an individualized dietary behavioural change (IDBC) programme and exercise training, in combination (COMB group) and separately (EXER-only and IDBC-only groups), to counteract sarcopenic obesity when compared with a control group receiving only health talks.
Who Masked: Outcomes Assessor
Masking Description: An independent assessor who is blinded to the group allocations will assess the participants' outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- The COMB group (Experimental): Participants in The COMB group will be grounded on the HAPA model and piloted by the team. It consists of three phases with 10 face-to-face hourly sessions nested with weekly telephone calls to enhance the participants' adherence to dietary behavioral change. And will be group-based, and offered weekly for about 60 minutes during the execution phase (a total 20 sessions from weeks 4-24). The combination of resistance and aerobic exercises can improve muscle quantity and strength as well as reduce body fat in people with sarcopenic obesity, and will be adopted in this study.
  Interventions: Behavioral: The Individualized Dietary Behavioural Change Programme (IDBC); Behavioral: The Exercise Training
- The EXER-only group (Experimental): Participants in The EXER-only group will be group-based, and offered weekly for about 60 minutes during the execution phase (a total 20 sessions from weeks 4-24). The combination of resistance and aerobic exercises can improve muscle quantity and strength as well as reduce body fat in people with sarcopenic obesity, and will be adopted in this study.
  Interventions: Behavioral: The Exercise Training
- The IDBC-only group (Experimental): Participants in The IDBC-only group will be grounded on the HAPA model and piloted by the team. It consists of three phases with 10 face-to-face hourly sessions nested with weekly telephone calls to enhance the participants' adherence to dietary behavioral change. And attend centre-based health talks about the management of different health issues with the exception of sarcopenic obesity.
  Interventions: Behavioral: The Individualized Dietary Behavioural Change Programme (IDBC)
- The Control Group (No Intervention): Participants in The Control Group will attend centre-based health talks about the management of different health issues with the exception of sarcopenic obesity. As the purpose of the health talk is to control the group interactive effect in exercise training, the group size, and the frequency and the time of the health talks will be similar to those offered in the exercise programme for the COMB and EXER-only groups.

INTERVENTIONS:
Behavioral: The Individualized Dietary Behavioural Change Programme (IDBC) — The first three weekly face-to-face sessions will be during the 'goal initiation' and 'planning' phases. The remaining seven face-to-face sessions will be offered once to twice per month between weeks 4 and 24 during the program at the 'action execution' phase. Family members will be encouraged to join the dietary consultations. Strategies will be discussed with the family members to facilitate the participant's adherence to the recommended diet regimen.Phase I Goal Initiation is aimed at motivating the participants to actively manage their sarcopenic obesity. Phase II Plan Formulation is aimed at guiding the participants in transforming their (sub-) goals into detailed individualized action plans.Phase III Action Execution is aimed at encouraging the participants to continually execute the action plan. The IDBC guidebook will be given to the participants to guide them on how to gradually adopt our dietary recommendations in their daily life.
  Arms: The COMB group; The IDBC-only group
Behavioral: The Exercise Training — The group size will be < 10. They will be used in the resistance exercise in this study to improve muscle strength (20 mins). Brisk walking (20 mins) will be employed in the aerobic exercise in this study. Each session will include 10 minutes of warm-up and cool-down exercises at the beginning and at the end. A YouTube video and a pamphlet describing the different types of exercises used in this programme will be disseminated to all participants to encourage them to continually practise their exercises at home for 30 minutes at least 5 times per week.
  Arms: The COMB group; The EXER-only group

SUMMARY:
Sarcopenic obesity (SO) has synergistic detrimental effects on elderlies' health. It greatly increases the risk of cardio-metabolic diseases, physical impairment, institutionalization, and mortality when compared with sarcopenia or obesity alone. Effective interventions to simultaneously increase muscle mass and decrease fat mass are challenging but highly warranted. Research showed that exercise tends to produce better outcomes in SO than nutritional interventions. Inconsistent effects of nutritional interventions may be due to a short intervention duration and participants' poor compliance with nutritional advice. Participants' adherence to a dietary regimen is essential to the success of nutritional interventions. Behavior change techniques grounded in a tested effective theoretical model - the Health Action Process Approach [HAPA] model at improving participants' self-efficacy should be incorporated in a diet modification intervention.This project aims to investigate the effects of a HAPA-based individualized dietary behavior change (IDBC) intervention and exercise training, in combination and separately, for elderly with SO, to improve their body composition and physical functions. In this four-armed randomized controlled trial, investigators will recruit and randomize 380 elderly with SO to one of the following four groups: the combined (COMB) group, receiving the 24-week combined intervention consisting of the IDBC program and exercise training, the EXER-only group, receiving only the exercise training, the IDBC-only group, receiving a combination of the IDBC program and health talks, and the control group, receiving only health talks with no other intervention. Investigators will use health talks to control the group and social interaction effects of the group exercise training for the COMB and the EXER-only groups. Investigators hypothesize that participants in the COMB, EXER-only, and IDBC-only groups will have significantly better outcome measures middle of the intervention (T1), immediately (T2), at 3-months (T3), and 6-months (T4) post-intervention than those in the control group when compared to baseline (T0).

Investigators will use mixed-effects modeling to compare changes in all outcome variables at the three post-tests among the four groups. If our intervention is effective at mitigating or preventing such occurrences, the impact on public health will be significant. A similar intervention for other populations.

DETAILED DESCRIPTION:
Low muscle mass and high body fat mass often coexist in older adults, a condition known as sarcopenic obesity. Older adults with low muscle mass and strength are 1.95-2.62 times more likely to suffer from obesity than those with normal muscle mass. This is because both sarcopenia and obesity have common risk factors that include unhealthy lifestyles and age-related physiological changes with a decline in growth hormones, increased insulin resistance, and increased oxidative stress. Sarcopenic obesity has synergistic detrimental effects on physical functions and overall health. The risks of developing cardio-metabolic diseases, institutionalization, and mortality are higher than with sarcopenia or obesity alone. Depending on the diagnostic criteria, its prevalence can be up to 20.4% and 27.0% in women and men, respectively, in China and worldwide.

Effective interventions to simultaneously increase muscle mass and decrease body fat mass are challenging, but highly warranted. To date, only a limited number of trials have focused on managing sarcopenic obesity. The common proposed interventions are lifestyle interventions (i.e. exercise and a nutritional intervention). Unfortunately, evidence-based interventions are yet to be established due to diverse methodologies with inconsistent results in different clinical trials.

Exercise-based interventions: The current evidence shows that managing sarcopenic obesity with exercise interventions tends to produce better outcomes than with nutritional interventions. A recent systematic review of 15 trials with 856 participants revealed that the combination of aerobic and resistance exercise decreased fat mass and improved physical performance (i.e. gait speed). However, additional benefits could not be observed when combining a nutritional intervention and exercise. Another systematic review of eight RCTs with 605 participants observed that resistance training alone could increase muscle strength. To also improve physical functions (i.e. gait speed and grip strength), exercise combining aerobic and resistance training with dietary supplements seems to have more promising results. Another systematic review of seven RCTs with 558 participants also reported that exercise alone or combined with dietary supplements showed beneficial effects on increasing muscle mass and physical functions in this population. In summary, exercise, especially the combination of resistance and aerobic training, improves body composition and physical performance in older adults with sarcopenic obesity. However, the additional beneficial effects of combining exercise and nutritional interventions were inconsistent.

Nutrition-based interventions: However, nutritional intervention should not be ignored in managing sarcopenic obesity, as unhealthy diet habit is a key factor to develop both sarcopenia (i.e. a result of an inadequate protein intake) and obesity (i.e. a result of an excess calories consumption). Studies suggest that adequate protein intake is essential for building muscles, whereas caloric restriction effectively reduces fat mass. Several studies demonstrated that a hypocaloric diet was effective in reducing fat mass in older adults with sarcopenic obesity. However, this fat mass loss is often accompanied with muscle mass loss. Therefore, a weight loss diet in this population should also focus on preserving muscle mass. Protein, particularly animal-based protein, which contains leucine, can prevent loss of muscle mass associated with weight reduction and maintain physical performance. Although dietary supplements are commonly used to increase protein intake, their effects on sarcopenic obesity remain inconsistent. Protein supplements may cause side effects, including dehydration, liver and renal damage, bloating, and calcium loss. Investigators argue that people should not only take dietary supplements but foods and meals containing a whole range of interacting constituents, which is also one of the points emphasized in the Dietary Guidelines for Americans, 2020-2025. Therefore, investigators believe that modifying the daily diet habits of people with sarcopenic obesity is more appropriate and may produce long-term benefits than solely giving them dietary supplements.

To date, only two intervention studies have attempted to modify the dietary habits of older adults with sarcopenic obesity. The first RCT compared the effects of a hypocaloric normal protein diet (0.8 g/kg body weight/day) and a hypocaloric high protein diet (1.2 g/kg body weight/day) for 3 months in 104 older women. The results showed a significant reduction in muscle mass associated with fat mass loss in the normal protein intake group, but increased muscle mass in the high protein group. This study provided preliminary evidence that a hypocaloric diet moderately rich in proteins was able to preserve muscle mass in their participants. Another pilot RCT found a significant reduction in muscle mass in a hypocaloric diet plus placebo group compared with a hypocaloric high-protein group (1.2-1.4 g / kg body weight / day) during a 4-month diet control regimen involving 18 women. The preliminary results showed that muscle strength improved significantly in the high-protein intake group, while no observable differences in fat free mass were observed in both groups. Some limitations were observed in these two studies, including the use of loose screening criteria for sarcopenic obesity without referring to a commonly accepted diagnostic standard, little information on the participants' compliance with the dietary regimen, and an unclear randomization process and intervention components. Further studies are required to examine the effects of using a diet modification approach on sarcopenic obesity in a rigorous manner.

The inconsistent effects of nutritional interventions may have been partly caused by a short intervention duration and/or poor adherence. A clinical trial found that muscle mass remained unchanged in the protein intake group until the nutritional programme had been implemented for 24 weeks. Hence, a longer duration (at least six months) is needed for a nutritional intervention to improve muscle mass-related parameters. Poor adherence and a high dropout rate were often reported in previous similar studies. A successful diet modification intervention requires improving the participants' adherence to the diet regimen. Therefore, behavioural change techniques grounded on a tested as effective theoretical model should be incorporated within a diet modification intervention.

Rationale for developing a dietary behavioural change programme grounded on the HAPA model: The Health Action Process Approach (HAPA) model divides the process of behavioural change into two phases: motivation and volition. The motivation phase refers to the goal initiation phase. 'Self-efficacy', 'outcome expectancies', and 'increased risk awareness' are the three attributes that motivate individuals to form an intention/goal to change their unhealthy lifestyle for a healthy lifestyle. The volition phase refers to the process of implementing intentions into actual behaviour through careful planning and action execution. The empirical evidence shows that the HAPA model can be effectively used as a conceptual framework to design concrete strategies to motivate behavioural changes. Used alongside dietary interventions, these strategies can promote adherence to diet advice on increasing fruit and vegetable consumption and to healthy dietary patterns and better nutritional behaviours.

Work done by the research team: Our team conducted a systematic review of 12 RCTs with 863 participants to identify evidence-based interventions for managing the problem. The results show that exercise, especially a combination of resistance and aerobic exercises, have better outcomes than nutritional inventions. This conclusion is similar to the findings in previous systematic reviews. Our meta-analysis showed that exercise combined with nutritional interventions significantly increased skeletal muscle mass when compared with the control group that received no intervention. With all the evidence, investigators believe nutritional interventions based on dietary modifications should be used for managing the problem. Investigators conducted a pilot two-armed RCT (Clinical Trial gov. NCT 04690985) on 60 older people with sarcopenic obesity to evaluate the feasibility and preliminary effects of an Individualized Dietary Behavioural Change (IDBC) programme. The design of the IDBC programme was grounded on a tested as effective HAPA model. The feasibility of the intervention was established by an acceptable recruitment rate (57.14%), a high retention rate (83.33%), and a high attendance rate (73.33% of participants attended five out of six dietary face-to-face consultation sessions). The participants did not report any adverse events. When compared with the control group, who received only health talks, participants in the IDBC group significantly reduced their body weight (IDBC vs Control=75.28kg to 74.78kg vs 72.29±1.40kg to 73.71±1.62kg, Wald χ2=4.90, p=0.027, d=1.22) and improved the quality of their diet (IDBC vs Control=60.03±2.02 to 65.92±2.35 vs 56.83±2.11 to 57.83±2.43, Wald χ2=12.66, p<0.001, d=1.31). Because it was a feasibility trial with insufficient power to identify significant changes, no significance difference could be identified in other outcome measurements. However, a trend of increased physical function (i.e., handgrip strength increased from [T1]:15.37±1.08 kg to [T2]:18.21±1.68 kg) and 6-m gait speed (increased from [T1]:0.91±0.02 m/s to [T2]:0.99±0.03 m/s) was observed only in the IDBC group. The use of behavioural change techniques enhanced the participants' adherence to the dietary regimen as evidenced by 66.67% of the participants adhering to the hypocaloric diet and the recommended daily protein intake, as measured by the protein score of the Dietary Quality Index (DQI). In summary, the findings from our pilot study showed that the IDBC programme is feasible. Preliminary positive effects showed that the dietary habits of older adults could be modified, leading to reduce sarcopenic obesity. In view of inconsistent results, it is also worth evaluating if any additional benefits can be observed with a combined IDBC programme with exercise in a well-design clinical trial.

The principal investigator (PI) JL and the Co-Is (CL, PK, JW) are adept at conducting intervention studies to manage frailty-related problems in older people or their caregivers. Another Co-I (SN), who is a physiotherapist academic, has conducted many RCTs using an activity-based lifestyle intervention for managing different problems in older adults. Our strength is in conducting intervention studies involving older adults in the community. Each of us has good connections with community partners, making subject recruitment feasible. The Co-Is have all contributed to developing and verifying the lifestyle intervention protocols used in the pilot study, and have worked closely with the PI to update and modify the protocols in the proposed study. LKH is a nutritionist academic and has already contributed to the proposed study by advising on the nutritional regimen in the protocol. He will work closely with the team to ensure the smooth implementation of the IDBC programme. PL provided the statistical expertise needed during the writing of the proposal and will employ these skills in analysing the data from the study.

ELIGIBILITY:
Inclusion Criteria:

1. community-dwelling older people aged > 65 years
2. who meet the diagnostic criteria of sarcopenic obesity according to the Asian Sarcopenia Working Group (ASWG)41 and the WHO definition of obesity for the Asian population, respectively: 2a) Early stage sarcopenia refers to the fulfillment of one of the following criteria: low handgrip strength < 28 kg for men and < 18 kg for women, low muscle quality as reflected by low appendicular skeletal muscle mass (ASM) /height squared < 7 kg/m2 for men and <5.7 kg/m2 for women, or low physical performance with a Short Physical Performance Battery (SPPB) score of < 9; 2b) Obesity refers to the fulfillment of one of the following criteria: BMI ≥ 23kg/m2 or waist circumference ≥ 90 cm in men and ≥ 80 cm in women, or percentage of body fat > 30%;
3. able to communicate, read, and write in Chinese without significant hearing and vision problems to ensure that our instructions are understood.

Exclusion Criteria:

1. those with any form of disease or condition that might affect food intake and digestion (such as severe heart or lung diseases, renal diseases, diabetes, cancer, or autoimmune diseases);
2. taking medications that may influence eating behaviour, digestion, or metabolism (such as weight loss medication);
3. being addicted to alcohol, which might affect the effort to change dietary behaviour;
4. having impaired mobility, which might affect participation in exercise training, as defined by a modified Functional Ambulatory Classification score of < 7; ) having any medical implant device such as a pacemaker, because low-level currents will flow through the body when doing the bioelectric impedance analysis (BIA by InBody s10, Korea), which may cause the device to malfunction.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Changes of muscle strength | Change from baseline to 12 weeks in the middle of the intervention, 24 weeks after the intervention, 3 months and 6 months after the programme
  Handgrip strength (kg) will be measured by using the jamar dynamometer.
Changes of muscle mass | Change from baseline to 12 weeks in the middle of the intervention, 24 weeks after the intervention, 3 months and 6 months after the programme
  Muscle mass (kg) will be measured by using bioelectrical impedance analysis.
The Short Physical Performance Battery (SPPB) scale | Change from baseline to 12 weeks in the middle of the intervention, 24 weeks after the intervention, 3 months and 6 months after the programme
  The Short Physical Performance Battery (SPPB) scale will be used to measure physical function, which is a well-established tool for monitoring function in older people, which contains three kinds of assessments: stand for 10 seconds with feet in 3 different positions, 3-meter or 4-meter walking speed test, and time to rise from a chair for five times. The scores of SPPB range from 0 (worst performance) to 12 (best performance).
  The unabbreviated scale title: The Short Physical Performance Battery (SPPB) scale The minimum and maximum values: 0, 10 Higher scores mean a better performance
Changes of body mass index | Change from baseline to 12 weeks in the middle of the intervention, 24 weeks after the intervention, 3 months and 6 months after the programme
  The weight and height will be combined to report BMI in kg/m^2.
Waist circumference | Change from baseline to 12 weeks in the middle of the intervention, 24 weeks after the intervention, 3 months and 6 months after the programme
  To estimate your potential disease risk is to measure your waist circumference. Excessive abdominal fat may be serious because it places you at greater risk for developing obesity-related conditions, such as Type 2 Diabetes, high blood pressure, and coronary artery disease.
Changes of fat mass | Change from baseline to 12 weeks in the middle of the intervention, 24 weeks after the intervention, 3 months and 6 months after the programme
  Fat mass (kg) will be measured by using bioelectrical impedance analysis.

SECONDARY OUTCOMES:
Mini Nutritional Assessment (MNA) Short-form | Change from baseline to 12 weeks in the middle of the intervention, 24 weeks after the intervention, 3 months and 6 months after the programme
  Participants' nutritional status will be assessed through the Mini Nutritional Assessment (MNA). It is a simple and quick tool for assessing older people who are malnourished or at risk of malnutrition. The MNA Short-form contains 6 items. Questions are weighted, 2-3 points per item. Scores are categorised as 0-7 (malnourished), 8-11 (at risk of malnutrition), 12-14 (normal nutritional status).
  The unabbreviated scale title: Mini Nutritional Assessment (MNA) Short-form The minimum and maximum values: 0, 14 Higher scores mean a better nutritional status
Diet Adherence | Change from baseline to 12 weeks in the middle of the intervention, 24 weeks after the intervention, 3 months and 6 months after the programme
  The adherence to protein intake will be reflected by the protein score in the DQI-I. Total calorie intake will be analyzed by a software program "Food Processor®". If any participant forgets to keep the dietary record, the 3-day food recall method will be used by the IDBC facilitator to check the participant's food intake, an approach commonly used in nutritional studies. The participants' attendance rate in the consultation sessions will be monitored.
Exercise Adherence | Change from baseline to 12 weeks in the middle of the intervention, 24 weeks after the intervention, 3 months and 6 months after the programme
  Assessed based on the participants' attendance in the weekly exercise training session, as well as on their self-reports on their overall adherence to the exercise regimen.
Health action process approach(HAPA)Nutrition Self-efficacy Scale | Change from baseline to 12 weeks in the middle of the intervention, 24 weeks after the intervention, 3 months and 6 months after the programme
  The nutrition self-efficacy scale is one part of the Health-Specific Self-efficacy Scale which was developed by Ralf Schwarzer and Britta Renner. The nutritional self-efficacy scale is a 5-item scale, and each item is rated on 4-point likert scale from 1= very uncertain, 2=rather uncertain, 3=rather certain, 4=very certain. Higher score means higher self-efficacy.
  The unabbreviated scale title: Health action process approach(HAPA)Nutrition Self-efficacy Scale The minimum and maximum values: 0, 20 Higher scores mean a higher self-efficacy
Dietary quality index-International (DQI-I) | Change from baseline to 12 weeks in the middle of the intervention, 24 weeks after the intervention, 3 months and 6 months after the programme
  The DQI-I will be used to estimate the dietary quality of participants. It is a well-used questionnaire without being affected by culture. The total scores range from 0 to 100, with a higher score representing better diet quality.
  The unabbreviated scale title: The Dietary quality index-International (DQI-I) The minimum and maximum values: 0, 100 Higher scores mean a better diet quality

CONTACTS AND LOCATIONS:
Overall Officials: Justina Liu, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
For confidentiality, the data will be kept anonymous and the information of all participants will be replaced by reference codes. The data collected will be kept in a locked place and electronic versions will be encrypted, and only be accessible by the researchers. All data will be destroyed within 7 years after the completion of this research.

REFERENCES:
- [Background] St-Onge MP, Gallagher D. Body composition changes with aging: the cause or the result of alterations in metabolic rate and macronutrient oxidation? Nutrition. 2010 Feb;26(2):152-5. doi: 10.1016/j.nut.2009.07.004. Epub 2009 Dec 8. PMID 20004080
- [Background] Kelley GA, Kelley KS. Is sarcopenia associated with an increased risk of all-cause mortality and functional disability? Exp Gerontol. 2017 Oct 1;96:100-103. doi: 10.1016/j.exger.2017.06.008. Epub 2017 Jun 21. PMID 28647519
- [Background] Brady AO, Straight CR, Evans EM. Body composition, muscle capacity, and physical function in older adults: an integrated conceptual model. J Aging Phys Act. 2014 Jul;22(3):441-52. doi: 10.1123/japa.2013-0009. Epub 2013 Aug 12. PMID 23945551
- [Background] Baumgartner RN, Wayne SJ, Waters DL, Janssen I, Gallagher D, Morley JE. Sarcopenic obesity predicts instrumental activities of daily living disability in the elderly. Obes Res. 2004 Dec;12(12):1995-2004. doi: 10.1038/oby.2004.250. PMID 15687401
- [Background] Prado CM, Wells JC, Smith SR, Stephan BC, Siervo M. Sarcopenic obesity: A Critical appraisal of the current evidence. Clin Nutr. 2012 Oct;31(5):583-601. doi: 10.1016/j.clnu.2012.06.010. Epub 2012 Jul 17. PMID 22809635
- [Background] Yin YH, Liu JYW, Valimaki M. Effectiveness of non-pharmacological interventions on the management of sarcopenic obesity: A systematic review and meta-analysis. Exp Gerontol. 2020 Jul 1;135:110937. doi: 10.1016/j.exger.2020.110937. Epub 2020 Mar 30. PMID 32240820
- [Background] Goisser S, Kemmler W, Porzel S, Volkert D, Sieber CC, Bollheimer LC, Freiberger E. Sarcopenic obesity and complex interventions with nutrition and exercise in community-dwelling older persons--a narrative review. Clin Interv Aging. 2015 Aug 6;10:1267-82. doi: 10.2147/CIA.S82454. eCollection 2015. PMID 26346071
- [Background] Katsanos CS, Kobayashi H, Sheffield-Moore M, Aarsland A, Wolfe RR. Aging is associated with diminished accretion of muscle proteins after the ingestion of a small bolus of essential amino acids. Am J Clin Nutr. 2005 Nov;82(5):1065-73. doi: 10.1093/ajcn/82.5.1065. PMID 16280440
- [Background] Mathus-Vliegen EM; Obesity Management Task Force of the European Association for the Study of Obesity. Prevalence, pathophysiology, health consequences and treatment options of obesity in the elderly: a guideline. Obes Facts. 2012;5(3):460-83. doi: 10.1159/000341193. Epub 2012 Jun 30. PMID 22797374
- [Background] Muscariello E, Nasti G, Siervo M, Di Maro M, Lapi D, D'Addio G, Colantuoni A. Dietary protein intake in sarcopenic obese older women. Clin Interv Aging. 2016 Feb 5;11:133-40. doi: 10.2147/CIA.S96017. eCollection 2016. PMID 26917955
- [Background] Sammarco R, Marra M, Di Guglielmo ML, Naccarato M, Contaldo F, Poggiogalle E, Donini LM, Pasanisi F. Evaluation of Hypocaloric Diet With Protein Supplementation in Middle-Aged Sarcopenic Obese Women: A Pilot Study. Obes Facts. 2017;10(3):160-167. doi: 10.1159/000468153. Epub 2017 May 20. PMID 28528340
- [Background] Newman AB, Lee JS, Visser M, Goodpaster BH, Kritchevsky SB, Tylavsky FA, Nevitt M, Harris TB. Weight change and the conservation of lean mass in old age: the Health, Aging and Body Composition Study. Am J Clin Nutr. 2005 Oct;82(4):872-8; quiz 915-6. doi: 10.1093/ajcn/82.4.872. PMID 16210719
- [Background] Stenholm S, Harris TB, Rantanen T, Visser M, Kritchevsky SB, Ferrucci L. Sarcopenic obesity: definition, cause and consequences. Curr Opin Clin Nutr Metab Care. 2008 Nov;11(6):693-700. doi: 10.1097/MCO.0b013e328312c37d. PMID 18827572
- [Background] Polyzos SA, Margioris AN. Sarcopenic obesity. Hormones (Athens). 2018 Sep;17(3):321-331. doi: 10.1007/s42000-018-0049-x. Epub 2018 Jul 16. PMID 30014320
- [Background] Kob R, Bollheimer LC, Bertsch T, Fellner C, Djukic M, Sieber CC, Fischer BE. Sarcopenic obesity: molecular clues to a better understanding of its pathogenesis? Biogerontology. 2015 Feb;16(1):15-29. doi: 10.1007/s10522-014-9539-7. Epub 2014 Nov 7. PMID 25376109
- [Background] Nakano R, Takebe N, Ono M, Hangai M, Nakagawa R, Yashiro S, Murai T, Nagasawa K, Takahashi Y, Satoh J, Ishigaki Y. Involvement of oxidative stress in atherosclerosis development in subjects with sarcopenic obesity. Obes Sci Pract. 2017 Jan 27;3(2):212-218. doi: 10.1002/osp4.97. eCollection 2017 Jun. PMID 28702214
- [Background] Godziuk K, Prado CM, Woodhouse LJ, Forhan M. The impact of sarcopenic obesity on knee and hip osteoarthritis: a scoping review. BMC Musculoskelet Disord. 2018 Jul 28;19(1):271. doi: 10.1186/s12891-018-2175-7. PMID 30055599
- [Background] Kim TN, Choi KM. The implications of sarcopenia and sarcopenic obesity on cardiometabolic disease. J Cell Biochem. 2015 Jul;116(7):1171-8. doi: 10.1002/jcb.25077. PMID 25545054
- [Background] Lim S, Kim JH, Yoon JW, Kang SM, Choi SH, Park YJ, Kim KW, Lim JY, Park KS, Jang HC. Sarcopenic obesity: prevalence and association with metabolic syndrome in the Korean Longitudinal Study on Health and Aging (KLoSHA). Diabetes Care. 2010 Jul;33(7):1652-4. doi: 10.2337/dc10-0107. Epub 2010 May 11. PMID 20460442
- [Background] Batsis JA, Mackenzie TA, Lopez-Jimenez F, Bartels SJ. Sarcopenia, sarcopenic obesity, and functional impairments in older adults: National Health and Nutrition Examination Surveys 1999-2004. Nutr Res. 2015 Dec;35(12):1031-9. doi: 10.1016/j.nutres.2015.09.003. Epub 2015 Sep 7. PMID 26472145
- [Background] Trouwborst I, Verreijen A, Memelink R, Massanet P, Boirie Y, Weijs P, Tieland M. Exercise and Nutrition Strategies to Counteract Sarcopenic Obesity. Nutrients. 2018 May 12;10(5):605. doi: 10.3390/nu10050605. PMID 29757230
- [Background] Hsu KJ, Liao CD, Tsai MW, Chen CN. Effects of Exercise and Nutritional Intervention on Body Composition, Metabolic Health, and Physical Performance in Adults with Sarcopenic Obesity: A Meta-Analysis. Nutrients. 2019 Sep 9;11(9):2163. doi: 10.3390/nu11092163. PMID 31505890
- [Background] Martinez-Amat A, Aibar-Almazan A, Fabrega-Cuadros R, Cruz-Diaz D, Jimenez-Garcia JD, Perez-Lopez FR, Achalandabaso A, Barranco-Zafra R, Hita-Contreras F. Exercise alone or combined with dietary supplements for sarcopenic obesity in community-dwelling older people: A systematic review of randomized controlled trials. Maturitas. 2018 Apr;110:92-103. doi: 10.1016/j.maturitas.2018.02.005. Epub 2018 Feb 13. PMID 29563041
- [Background] Hita-Contreras F, Bueno-Notivol J, Martinez-Amat A, Cruz-Diaz D, Hernandez AV, Perez-Lopez FR. Effect of exercise alone or combined with dietary supplements on anthropometric and physical performance measures in community-dwelling elderly people with sarcopenic obesity: A meta-analysis of randomized controlled trials. Maturitas. 2018 Oct;116:24-35. doi: 10.1016/j.maturitas.2018.07.007. Epub 2018 Jul 19. PMID 30244776
- [Background] McCarthy D, Berg A. Weight Loss Strategies and the Risk of Skeletal Muscle Mass Loss. Nutrients. 2021 Jul 20;13(7):2473. doi: 10.3390/nu13072473. PMID 34371981
- [Background] Anthony TG. Mechanisms of protein balance in skeletal muscle. Domest Anim Endocrinol. 2016 Jul;56 Suppl(Suppl):S23-32. doi: 10.1016/j.domaniend.2016.02.012. PMID 27345321
- [Background] Bauer J, Biolo G, Cederholm T, Cesari M, Cruz-Jentoft AJ, Morley JE, Phillips S, Sieber C, Stehle P, Teta D, Visvanathan R, Volpi E, Boirie Y. Evidence-based recommendations for optimal dietary protein intake in older people: a position paper from the PROT-AGE Study Group. J Am Med Dir Assoc. 2013 Aug;14(8):542-59. doi: 10.1016/j.jamda.2013.05.021. Epub 2013 Jul 16. PMID 23867520
- [Background] Schaafsma G. Safety of protein hydrolysates, fractions thereof and bioactive peptides in human nutrition. Eur J Clin Nutr. 2009 Oct;63(10):1161-8. doi: 10.1038/ejcn.2009.56. Epub 2009 Jul 22. PMID 19623200
- [Background] Wolfe RR. Protein supplements and exercise. Am J Clin Nutr. 2000 Aug;72(2 Suppl):551S-7S. doi: 10.1093/ajcn/72.2.551S. PMID 10919959
- [Background] Desroches S, Lapointe A, Ratte S, Gravel K, Legare F, Turcotte S. Interventions to enhance adherence to dietary advice for preventing and managing chronic diseases in adults. Cochrane Database Syst Rev. 2013 Feb 28;2013(2):CD008722. doi: 10.1002/14651858.CD008722.pub2. PMID 23450587
- [Background] Zhou X, Xing B, He G, Lyu X, Zeng Y. The Effects of Electrical Acupuncture and Essential Amino Acid Supplementation on Sarcopenic Obesity in Male Older Adults: A Randomized Control Study. Obes Facts. 2018;11(4):327-334. doi: 10.1159/000491797. Epub 2018 Aug 9. PMID 30089292
- [Background] Burgess E, Hassmen P, Pumpa KL. Determinants of adherence to lifestyle intervention in adults with obesity: a systematic review. Clin Obes. 2017 Jun;7(3):123-135. doi: 10.1111/cob.12183. Epub 2017 Mar 15. PMID 28296261
- [Background] Schwarzer R, Warner LM, Fleig L, Gholami M, Serra-Majem L, Ngo J, Cianferotti L, Kritikou M, Mossi P, Ntzani E, Brandi ML. Dietary planning, self-efficacy, and outcome expectancies play a role in an online intervention on fruit and vegetable consumption. Psychol Health. 2018 May;33(5):652-668. doi: 10.1080/08870446.2017.1385785. Epub 2017 Oct 9. PMID 28990404
- [Background] Schwarzer R, Renner B. Social-cognitive predictors of health behavior: action self-efficacy and coping self-efficacy. Health Psychol. 2000 Sep;19(5):487-95. PMID 11007157
- [Background] Chen LK, Liu LK, Woo J, Assantachai P, Auyeung TW, Bahyah KS, Chou MY, Chen LY, Hsu PS, Krairit O, Lee JS, Lee WJ, Lee Y, Liang CK, Limpawattana P, Lin CS, Peng LN, Satake S, Suzuki T, Won CW, Wu CH, Wu SN, Zhang T, Zeng P, Akishita M, Arai H. Sarcopenia in Asia: consensus report of the Asian Working Group for Sarcopenia. J Am Med Dir Assoc. 2014 Feb;15(2):95-101. doi: 10.1016/j.jamda.2013.11.025. PMID 24461239
- [Background] Pavasini R, Guralnik J, Brown JC, di Bari M, Cesari M, Landi F, Vaes B, Legrand D, Verghese J, Wang C, Stenholm S, Ferrucci L, Lai JC, Bartes AA, Espaulella J, Ferrer M, Lim JY, Ensrud KE, Cawthon P, Turusheva A, Frolova E, Rolland Y, Lauwers V, Corsonello A, Kirk GD, Ferrari R, Volpato S, Campo G. Short Physical Performance Battery and all-cause mortality: systematic review and meta-analysis. BMC Med. 2016 Dec 22;14(1):215. doi: 10.1186/s12916-016-0763-7. PMID 28003033
- [Background] Liu P, Ma F, Lou H, Zhu Y. Utility of obesity indices in screening Chinese postmenopausal women for metabolic syndrome. Menopause. 2014 May;21(5):509-14. doi: 10.1097/GME.0b013e3182a170be. PMID 23963310
- [Background] Kraus WE, Bhapkar M, Huffman KM, Pieper CF, Krupa Das S, Redman LM, Villareal DT, Rochon J, Roberts SB, Ravussin E, Holloszy JO, Fontana L; CALERIE Investigators. 2 years of calorie restriction and cardiometabolic risk (CALERIE): exploratory outcomes of a multicentre, phase 2, randomised controlled trial. Lancet Diabetes Endocrinol. 2019 Sep;7(9):673-683. doi: 10.1016/S2213-8587(19)30151-2. Epub 2019 Jul 11. PMID 31303390
- [Background] Tome D. Muscle Protein Synthesis and Muscle Mass in Healthy Older Men. J Nutr. 2017 Dec;147(12):2209-2211. doi: 10.3945/jn.117.263491. Epub 2017 Nov 1. No abstract available. PMID 29093015
- [Background] Deutz NE, Bauer JM, Barazzoni R, Biolo G, Boirie Y, Bosy-Westphal A, Cederholm T, Cruz-Jentoft A, Krznaric Z, Nair KS, Singer P, Teta D, Tipton K, Calder PC. Protein intake and exercise for optimal muscle function with aging: recommendations from the ESPEN Expert Group. Clin Nutr. 2014 Dec;33(6):929-36. doi: 10.1016/j.clnu.2014.04.007. Epub 2014 Apr 24. PMID 24814383
- [Background] Morley JE, Argiles JM, Evans WJ, Bhasin S, Cella D, Deutz NE, Doehner W, Fearon KC, Ferrucci L, Hellerstein MK, Kalantar-Zadeh K, Lochs H, MacDonald N, Mulligan K, Muscaritoli M, Ponikowski P, Posthauer ME, Rossi Fanelli F, Schambelan M, Schols AM, Schuster MW, Anker SD; Society for Sarcopenia, Cachexia, and Wasting Disease. Nutritional recommendations for the management of sarcopenia. J Am Med Dir Assoc. 2010 Jul;11(6):391-6. doi: 10.1016/j.jamda.2010.04.014. PMID 20627179
- [Background] Paddon-Jones D, Leidy H. Dietary protein and muscle in older persons. Curr Opin Clin Nutr Metab Care. 2014 Jan;17(1):5-11. doi: 10.1097/MCO.0000000000000011. PMID 24310053
- [Background] Eyles HC, Mhurchu CN. Does tailoring make a difference? A systematic review of the long-term effectiveness of tailored nutrition education for adults. Nutr Rev. 2009 Aug;67(8):464-80. doi: 10.1111/j.1753-4887.2009.00219.x. PMID 19674343
- [Background] Kim H, Kim M, Kojima N, Fujino K, Hosoi E, Kobayashi H, Somekawa S, Niki Y, Yamashiro Y, Yoshida H. Exercise and Nutritional Supplementation on Community-Dwelling Elderly Japanese Women With Sarcopenic Obesity: A Randomized Controlled Trial. J Am Med Dir Assoc. 2016 Nov 1;17(11):1011-1019. doi: 10.1016/j.jamda.2016.06.016. Epub 2016 Aug 17. PMID 27544583
- [Background] Liao CD, Tsauo JY, Huang SW, Ku JW, Hsiao DJ, Liou TH. Effects of elastic band exercise on lean mass and physical capacity in older women with sarcopenic obesity: A randomized controlled trial. Sci Rep. 2018 Feb 2;8(1):2317. doi: 10.1038/s41598-018-20677-7. PMID 29396436
- [Background] Park J, Kwon Y, Park H. Effects of 24-Week Aerobic and Resistance Training on Carotid Artery Intima-Media Thickness and Flow Velocity in Elderly Women with Sarcopenic Obesity. J Atheroscler Thromb. 2017 Nov 1;24(11):1117-1124. doi: 10.5551/jat.39065. Epub 2017 Jul 1. PMID 28674320
- [Background] Bird EL, Baker G, Mutrie N, Ogilvie D, Sahlqvist S, Powell J. Behavior change techniques used to promote walking and cycling: a systematic review. Health Psychol. 2013 Aug;32(8):829-38. doi: 10.1037/a0032078. Epub 2013 Mar 11. PMID 23477577
- [Background] Guerra RS, Amaral TF. Comparison of hand dynamometers in elderly people. J Nutr Health Aging. 2009 Dec;13(10):907-12. doi: 10.1007/s12603-009-0250-3. PMID 19924352
- [Background] Zhou G, Jiang T, Knoll N, Schwarzer R. Improving hand hygiene behaviour among adolescents by a planning intervention. Psychol Health Med. 2015;20(7):824-31. doi: 10.1080/13548506.2015.1024138. Epub 2015 Mar 16. PMID 25774807
- [Background] Woo J, Cheung B, Ho S, Sham A, Lam TH. Influence of dietary pattern on the development of overweight in a Chinese population. Eur J Clin Nutr. 2008 Apr;62(4):480-7. doi: 10.1038/sj.ejcn.1602702. Epub 2007 Feb 28. PMID 17327865
- [Background] Kim S, Haines PS, Siega-Riz AM, Popkin BM. The Diet Quality Index-International (DQI-I) provides an effective tool for cross-national comparison of diet quality as illustrated by China and the United States. J Nutr. 2003 Nov;133(11):3476-84. doi: 10.1093/jn/133.11.3476. PMID 14608061
- [Background] Yang YJ, Kim MK, Hwang SH, Ahn Y, Shim JE, Kim DH. Relative validities of 3-day food records and the food frequency questionnaire. Nutr Res Pract. 2010 Apr;4(2):142-8. doi: 10.4162/nrp.2010.4.2.142. Epub 2010 Apr 28. PMID 20461203
- [Background] Kreidler SM, Muller KE, Grunwald GK, Ringham BM, Coker-Dukowitz ZT, Sakhadeo UR, Baron AE, Glueck DH. GLIMMPSE: Online Power Computation for Linear Models with and without a Baseline Covariate. J Stat Softw. 2013 Sep;54(10):i10. doi: 10.18637/jss.v054.i10. PMID 24403868
- [Background] Bellg AJ, Borrelli B, Resnick B, Hecht J, Minicucci DS, Ory M, Ogedegbe G, Orwig D, Ernst D, Czajkowski S; Treatment Fidelity Workgroup of the NIH Behavior Change Consortium. Enhancing treatment fidelity in health behavior change studies: best practices and recommendations from the NIH Behavior Change Consortium. Health Psychol. 2004 Sep;23(5):443-51. doi: 10.1037/0278-6133.23.5.443. PMID 15367063
- See also: Dietary Guidelines for Americans, 2020-2025 — http://www.dietaryguidelines.gov/sites/default/files/2020-12/Dietary_Guidelines_for_Americans_2020-2025.pdf
- See also: The Asia-Pacific perspective: redefining obesity and its treatment — http://apps.who.int/iris/handle/10665/206936
- See also: Centre for Health Protection Hong Kong. Obesity: A Weighty Health Issue Key Messages — http://www.chp.gov.hk/files/pdf/ncd_watch_august_2018.pdf
- See also: Research E. Food Processor® software — http://www.esha.com

DOCUMENTS (1):
  • Informed Consent Form (2023-02-10): https://cdn.clinicaltrials.gov/large-docs/55/NCT05734755/ICF_000.pdf